CLINICAL TRIAL: NCT05021861
Title: Evaluation of Periodontal Status and High Sensitivity C Reactive Protein Levels in Female Patients Diagnosed With Polycystic Ovary Syndrome on Cyproterone Acetate/Ethinyl Estradiol Combination Regimen: a Cross Sectional Study
Brief Title: Evaluation of Periodontal Status and hsCRP Levels in Females With PCOS on CPA/EE Combination Drug Regimen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: RidhimaPerio
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis; Polycystic Ovary Syndrome; Gingivitis
MeSH Terms: conditions — Periodontitis; Polycystic Ovary Syndrome; Gingivitis | interventions — Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Test group 1: FEMALE PATIENTS WITH PCOS ON CPA/EE DRUG REGIMEN FOR ATLEAST 6 MONTHS.
  Interventions: Drug: Cyproterone Acetate, Ethinyl Estradiol Drug Combination
- Test group 2: FEMALE PATIENTS WITH PCOS( NEWLY DIAGNOSED) ,NOT ON ANY MEDICATION,
  Interventions: Diagnostic Test: FEMALE PATIENTS WITH PCOS
- Control group: SYSTEMICALLY HEALTHY FEMALES
  Interventions: Diagnostic Test: Control group

INTERVENTIONS:
Drug: Cyproterone Acetate, Ethinyl Estradiol Drug Combination — FEMALE PATIENTS WITH PCOS ON CPA/EE DRUG REGIMEN FOR ATLEAST 6 MONTHS
  Other Names: Diane-35
  Groups: Test group 1
Diagnostic Test: FEMALE PATIENTS WITH PCOS — FEMALE PATIENTS WITH PCOS( NEWLY DIAGNOSED) ,NOT ON ANY MEDICATION,
  Groups: Test group 2
Diagnostic Test: Control group — SYSTEMICALLY HEALTHY FEMALES
  Groups: Control group

SUMMARY:
PCOS is a widely reported condition among young female population and anti-androgen agents are increasingly being used as part of the medical management of such cases. However, Clinical studies have reported higher prevalence of gingival inflammation, loss of attachment and gingival enlargement in women taking hormone based oral contraceptives. Additionally, CPA has been reported to have an osteoclastic action. Therefore, it is necessary to explore whether these medications affect the periodontal condition of PCOS patients, who already are pre-disposed to systemic inflammation. Therefore, the present study aims to evaluate the periodontal status of female patients diagnosed with Polycystic Ovary syndrome on Cyproterone acetate/ethinyl estradiol combination regimen.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a complex endocrine, reproductive and metabolic condition, affecting women of reproductive age globally with a worldwide prevalence ranging from 5-15%.It is characterised by elevation of multiple markers of inflammation such as C-reactive protein (CRP), proinflammatory cytokines and chemokines, white blood cell count as well as increased oxidative stress.

It has been hypothesised that PCOS might exacerbate the periodontal condition that is caused by dental plaque, through various pathophysiological links, namely, low-grade systemic inflammation, oxidative stress, insulin resistance (IR), advanced glycation end products (AGE), and systemic hormonal levels. Evidence has suggested that periodontal disease causes chronic subclinical inflammation leading to Insulin resistance, initiating the development of type 2 diabetes, which in turn is a prominent feature in PCOS. Hence, a two-way relationship between PCOS and periodontal disease is currently being explored There exists a pathological imbalance of Luteinizing Hormone(LH) and Follicle Stimulating Hormone (FSH) in women with PCOS which explains the rationale for treatment with combined hormonal treatment.11 These treatments include combined oral contraceptives (COCs) and anti androgen tharapy (ADT) in the form of antiandrogenic progestogen/ ethinylestradiol (EE) combinations.

Receptors for estrogen have been demonstrated in the gingiva and periodontal connective tissue cells While the effects of different contraceptive combinations and/or oral hypoglycemics on the periodontal condition of female patients diagnosed with PCOS has been explored, the specific drug combination of CPA/EE has not been studied in detail as yet.

The present study aims to evaluate the periodontal status of female patients diagnosed with PCOS on CPA/EE combination regimen.

MATERIALS AND METHODS- The present cross-sectional study will be conducted in the Department of periodontology, Post Graduate Institute of Dental Sciences, Rohtak in collaboration with Department of Obstetrics and Gynaecology Post Graduate Institute of Medical Sciences, Rohtak over a period of 12-14 months in Female patients diagnosed with PCOS.It will include 150 individuals, who will be comprised into 3 groups and the individuals in each group will be recruited as Test group 1- Female patients diagnosed with PCOS ON CPA/EE DRUG REGIMEN FOR ATLEAST 6 MONTHS.

Test group 2- Female patients diagnosed with PCOS( NEWLY DIAGNOSED) ,NOT ON ANY MEDICATION, Control group -SYSTEMICALLY HEALTHY FEMALES

The primary outcome measures include bleeding on probing (BOP),Probing pocket depth(PPD),Clinical attachment level(CAL),Serum High Sensitivity C- reactive Proteins (hsCRP).SECONDARY MEASURES include Plaque index, Gingival index,Gingival phenotype,Gingival recession,Demographic parameters ( Education status, Socio-economic status),Anthropometric parameters (Waist circumference, waist to hip ratio, Body mass index) ,Quality of life ( via PCOS Questionnaire, Oral health related Questionnaire).

DATA MANAGEMENT AND STATISTICAL ANALYSIS - Data recorded will be processed by standard statistical analysis.The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution inter group comparison will be done by using Independent T test between signed rank test and if in non-normal distribution inter group comparison will be done by Mann-Whitney U test. The Chi square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females of age group (15-40yrs) diagnosed with PCOS. The diagnosis of PCOS will be according to Rotterdam criteria, when any two out of the following three abnormalities will be present:

  1. clinical (hirsutism, acne or acanthosis nigricans) and/or biochemical (raised testosterone) hyperandrogenism ;
  2. chronic anovulation (oligomenorrhoea or amenorrhea); and
  3. polycystic ovaries on ultrasound (one or both ovaries demonstrate 12 or more follicles measuring 2 to 9 mm in diameter or the ovarian volume exceeds 10 cubic cm on pelvic ultrasound) from department of Obstetrics and Gynaecology, Post Graduate Institute of Medical Sciences, Rohtak.
* presence of ≥20 natural teeth
* BMI (18.5 - 24.9)
* Systemically healthy females {Age and BMI matched with PCOS women} diagnosed on the basis of

  1. Regular mensturation,
  2. No clinical or biochemical sign of hyperandrogenism and
  3. Ultrasound exclusion of PCOS

Exclusion Criteria:

* Previous history of androgen-secreting tumors, congenital adrenal hyperplasia , hyperprolactinemia, or any thyroid dysfunction
* Patients with chronic inflammatory disease such as nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, or active cancer within the past 5 years
* Smokers and alcoholics,
* History of systemic antibiotics or oral contraceptives usage within last 3 months,
* Periapical pathology or other oral inflammatory conditions and any periodontal treatment within 6 months prior to study

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — self-representation of gender identity
Study Population: Female patients diagnosed with PCOS on CPA/EE combination drug regimen.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing | 6 months
  Percentage of bleeding sites on probing
Pocket depth | 6 months
  Distance from gingival margin to base of the pocket
HsCRP levels | 6 months
  C reactive protein levels in serum

CONTACTS AND LOCATIONS:
Overall Officials: RIDHIMA SINGHAL, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India